CLINICAL TRIAL: NCT03182218
Title: Prospective Observational Study of the Direct Oral Anticoagulants Periprocedural Management
Brief Title: Periprocedural Direct Oral Anticoagulant Management
Acronym: RA-ACOD
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Raquel Ferrandis, Doctor, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: INC-ACO-2013-01
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Periprocedural Complication
Keywords: Periprocedural; Anticoagulation; Dabigatran; Rivaroxaban; Apixaban; Edoxaban; Direct oral anticoagulant; Surgery; Anaesthesia; Novel oral anticoagulant; Perioperative medicine
MeSH Terms: interventions — N(4)-oleylcytosine arabinoside; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Direct oral anticoagulant — Time of direct oral anticoagulant withdrawal Use or not of bridging with low molecular weight heparin
  Other Names: low molecular weight heparin

SUMMARY:
Direct oral anticoagulants (DOAC) are a new drug group that has been approved for chronic anticoagulation of patients in atrial fibrillation or suffering acute thrombosis, between others. The need of surgery of a patient in atrial fibrillation is round 10% per year.

Due to DOAC short time of commercialization and the lack of experience, the proper management of DOAC when a patient in this treatment needs a scheduled or urgent procedure, has not yet been established. This fact may mean both the decrease of the anticoagulant treatment efficacy and the increase of the haemorrhage complications in the perioperative period.

With the aim of gaining additional information about this aspect, a multicentre, prospective and observational study (classified by the spanish drug society, AEMPS, as non-interventional trial, EPA-SP) about the DOAC management, before a scheduled or urgent surgery, in normal clinical practice, is proposed.

DETAILED DESCRIPTION:
When an anticoagulated patient is scheduled for surgery or an invasive procedure, the physician's worry is how to achieve needing an optimal haemostasis without increasing the risk of thrombosis. For decades, the main drug for chronic anticoagulation has been antivitamin-k (warfarin or acenocoumarol). In the majority of patients, the periprocedural management proposal has been stopping the drug and giving a short acting anticoagulant for some days before surgery, known as bridging therapy strategy, mostly done with a low-molecular weight heparin (LMWH).

The debate about the best perioperative management of the anticoagulated patients has increased with the arrival on the market of direct oral anticoagulants (DOAC), by the moment approved for long-term anticoagulation in patients with atrial fibrillation and for the treatment of pulmonary embolism. DOAC could be classified in two groups: direct inhibitors of thrombin (the only current available drug is dabigatran) and direct inhibitors of factor Xa (rivaroxaban, apixaban, edoxaban, and others soon to come). DOAC have pharmacokinetic characteristics that seem to favour stopping the drug for some days without substitution in the vast majority of the patients. Nevertheless, current lack of experience in the management of high doses of DOAC during the perioperative period, the absence of effective antagonists to reverse the anticoagulation, the unsuitable standardized laboratory monitoring and, also, the different pharmacokinetics between patients receiving these drugs, have made challenging to standardize the optimal management in the perioperative period. Some proposals have been published in last years from expert consensus, based on pharmacokinetic data, but DOAC short time of commercialization and the difficulties to interpret the post-hoc analysis from the randomized trials, for the heterogeneity of the included population and the wide kind of surgeries, most of them with low bleeding risk, have moved the spanish working group on perioperative management of haemostasis to plan a multi-institutional registry to gain experience and information in the periprocedural (urgent or scheduled) management of DOAC.

The authors designed an observational, prospective, multicentre study including patients under long-term DOAC treatment for atrial fibrillation or treatment of venous thromboembolism who are scheduled or need an urgent procedure. Data collected were demographic, related with the DOAC management and with the possible haemorrhagic or thrombotic events with a follow-up of 30 day. A univariable analysis and a multivariate regression model were applied using all the available co-variables. Bilateral hypothesis contrast were considered significant if α < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and older
* Under direct oral anticoagulant
* Urgent or scheduled surgery or invasive procedure needed
* Signed and dated informed consent form

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient under treatment with direct oral anticoagulant who requires a surgery or an invasive procedural, both scheduled or urgent.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Periprocedural thrombotic complications | 1 month
  Accumulative incidence rate of thrombotic events (cardiovascular, neurological, or venous thromboembolic event)
Periprocedural hemorrhagic complications | 1 month
  Accumulative incidence rate of minor and major bleeding events

SECONDARY OUTCOMES:
Outcome of bridging therapy | Between one week before and one month after procedural
  Relationship between the incidence of complications and the use of bridging therapy.
Knowing actual DOAC management in clinical practice | Between one week before and one month after procedural
  Composite of time of withdrawal of direct oral anticoagulant, use or not of low molecular weight heparin as bridge therapy, time of reintroduction of direct oral anticoagulant

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Ferrandis Comes, Doctor, Principal Investigator — Fundación para la Investigación del Hospital Clínico de Valencia
Locations (30):
- Spain (30):
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital de Sabadell-Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital de Manises, Manises, Valencia
  - Hospital Universitario La Ribera, Alzira
  - Parc Salut Mar, Barcelona
  - Fundació Puigvert, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital de Galdakao-Usánsolo, Galdakao
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Costa del Sol, Marbella
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario de Móstoles, Móstoles
  - Clínica Universidad de Navarra, Pamplona
  - Hospital General de Segovia, Segovia
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario, Valencia
  - Consorcio H. General Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Dr Peset, Valencia
  - Hospital Lluís Alcanyís, Xàtiva
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

REFERENCES:
- [Background] Perez-Villacastin J, Perez Castellano N, Moreno Planas J. Epidemiology of atrial fibrillation in Spain in the past 20 years. Rev Esp Cardiol (Engl Ed). 2013 Jul;66(7):561-5. doi: 10.1016/j.rec.2013.02.012. Epub 2013 May 28. PMID 24776206
- [Background] Barrios V, Calderon A, Escobar C, de la Figuera M; Primary Care Group in the Clinical Cardiology Section of the Spanish Society of Cardiology. Patients with atrial fibrillation in a primary care setting: Val-FAAP study. Rev Esp Cardiol (Engl Ed). 2012 Jan;65(1):47-53. doi: 10.1016/j.recesp.2011.08.008. Epub 2011 Nov 4. English, Spanish. PMID 22054913
- [Background] Cea-Calvo L, Redon J, Marti-Canales JC, Lozano JV, Llisterri JL, Fernandez-Perez C, Aznar J, Gonzalez-Esteban J. [Prevalence of low glomerular filtration rate in the elderly population of Spain. The PREV-ICTUS study]. Med Clin (Barc). 2007 Nov 17;129(18):681-7. doi: 10.1157/13112509. Spanish. PMID 18021608
- [Background] Weitz JI, Eikelboom JW, Samama MM. New antithrombotic drugs: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e120S-e151S. doi: 10.1378/chest.11-2294. PMID 22315258
- [Background] Wittkowsky AK. Novel oral anticoagulants and their role in clinical practice. Pharmacotherapy. 2011 Dec;31(12):1175-91. doi: 10.1592/phco.31.12.1175. PMID 22122180
- [Background] Mavrakanas T, Bounameaux H. The potential role of new oral anticoagulants in the prevention and treatment of thromboembolism. Pharmacol Ther. 2011 Apr;130(1):46-58. doi: 10.1016/j.pharmthera.2010.12.007. Epub 2010 Dec 24. PMID 21185864
- [Background] Llau JV, Ferrandis R, Castillo J, de Andres J, Gomar C, Gomez-Luque A, Hidalgo F, Torres LM. [Recommendations on use of direct oral anticoagulants in the perioperative period]. Med Clin (Barc). 2012 Oct;139 Suppl 2:46-50. doi: 10.1016/S0025-7753(12)70042-8. Spanish. PMID 23498073
- [Background] van Ryn J, Stangier J, Haertter S, Liesenfeld KH, Wienen W, Feuring M, Clemens A. Dabigatran etexilate--a novel, reversible, oral direct thrombin inhibitor: interpretation of coagulation assays and reversal of anticoagulant activity. Thromb Haemost. 2010 Jun;103(6):1116-27. doi: 10.1160/TH09-11-0758. Epub 2010 Mar 29. PMID 20352166
- [Background] Turpie AG, Kreutz R, Llau J, Norrving B, Haas S. Management consensus guidance for the use of rivaroxaban--an oral, direct factor Xa inhibitor. Thromb Haemost. 2012 Nov;108(5):876-86. doi: 10.1160/TH12-03-0209. Epub 2012 Sep 26. PMID 23014816
- [Background] Schulman S, Crowther MA. How I treat with anticoagulants in 2012: new and old anticoagulants, and when and how to switch. Blood. 2012 Mar 29;119(13):3016-23. doi: 10.1182/blood-2011-10-378950. Epub 2012 Feb 1. PMID 22302737
- [Background] Gallego P, Apostolakis S, Lip GY. Bridging evidence-based practice and practice-based evidence in periprocedural anticoagulation. Circulation. 2012 Sep 25;126(13):1573-6. doi: 10.1161/CIRCULATIONAHA.112.135681. No abstract available. PMID 23008469
- [Background] Llau JV, Ferrandis R. Letter by Llau and Ferrandis regarding article, "Bridging evidence-based practice and practice-based evidence in periprocedural anticoagulation". Circulation. 2013 May 14;127(19):e616. doi: 10.1161/CIRCULATIONAHA.112.151506. No abstract available. PMID 23671184
- [Background] Ferrandis R, Castillo J, de Andres J, Gomar C, Gomez-Luque A, Hidalgo F, Llau JV, Sierra P, Torres LM. The perioperative management of new direct oral anticoagulants: a question without answers. Thromb Haemost. 2013 Sep;110(3):515-22. doi: 10.1160/TH12-11-0868. Epub 2013 Jul 11. PMID 23846475